CLINICAL TRIAL: NCT05089487
Title: The Impact of Hypoxia on Patients With Precapillary Pulmonary Hypertension and Treatment of Adverse Effects
Brief Title: Nocturnal Oxygenation and Sleep-related Breathing Disorders During the First Night of a Stay at 2500m of High Altitude in Patients With Precapillary Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: OVERALP II E
Record Dates: First submitted 2021-10-14; First posted 2021-10-22 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: High Altitude Pulmonary Hypertension; Sleep
MeSH Terms: conditions — Pulmonary edema of mountaineers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High altitude 2500 m above sea level (Experimental)
  Interventions: Procedure: Nocturnal rest (sleep study)
- Low altitude 470 m above sea level (Active Comparator)
  Interventions: Procedure: Nocturnal rest (sleep study)

INTERVENTIONS:
Procedure: Nocturnal rest (sleep study) — Proportion of patients free of severe hypoxemia without oxygen therapy during nocturnal rest .

SUMMARY:
The impact of hypoxia at 2500m of high altitude on sleep in patients with precapillary pulmonary hypertension

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature (Appendix Informed Consent Form)
* PH class I (PAH) or IV (CTEPH) diagnosed according to guidelines: mean pulmonary artery pressure >20 mmHg, pulmonary vascular resistance ≥3 wood units, pulmonary arterial wedge pressure ≤15 mmHg during baseline measures at the diagnostic right-heart catheterization

Exclusion Criteria:

* resting partial pressure of oxygen <8 kilopascal at Zurich at 490 m low altitude
* exposure to an altitude >1000 m for ≥3 nights during the last 2 weeks before the study
* inability to follow the procedures of the study
* other clinically significant concomitant end-stage disease (e.g., renal failure, hepatic dysfunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients free of severe hypoxemia | 30 hours
  Proportion of patients free of severe hypoxemia (defined as oxygenation (SpO2)<80% for >30 min) without oxygen therapy during nocturnal rest at 2500 m vs. 490 m

SECONDARY OUTCOMES:
Nocturnal oxygenation | 30 hours
  Difference in mean nocturnal oxygenation (SpO2) 2500 m of high altitude vs 490 m low altitude
Oxygen desaturation index | 30 hours
  Difference in oxygen desaturation index sleeping at 2500 m high altitude vs 490 m low altitude
Periodic breathing | 30 hours
  Difference in time spent with periodic breathing in patients sleeping at 2500 m of high altitude vs 490 m low altitude
Nocturnal transcutaneous carbon dioxide tension | 30 hours
  Difference in nocturnal transcutaneous carbon dioxide tension in patients sleeping at 2500 m of high altitude vs 490 m low altitude
Visual Analogue Scale | 30 hours
  Subjective sleep quality Visual Analogue Scale score 2500 m high altitude vs 490 m low altitude
Time spent awake during the night | 30 hours
  Subjective time spent awake during the night high altitude vs 490 m low altitude
Cerebral tissue deoxygenation | 30 hours
  Proportion of patients free of severe cerebral tissue deoxygenation (drop in cerebral tissue oxygen saturation >5%) without oxygen therapy during a night at 2500 vs. 490 m
Cerebral tissue oxygen saturation awake | 30 hours
  Difference in cerebral tissue oxygen saturation awake in patients with precapillary pulmonary hypertension at 2500m of high altitude without supplemental oxygen vs. low altitude
Cerebral tissue oxygen saturation during sleep without oxygen | 30 hours
  Difference in cerebral tissue oxygen saturation during sleep in patients with precapillary pulmonary hypertension at 2500m of high altitude without supplemental oxygen
Cerebral tissue oxygen saturation during sleep with oxygen | 30 hours
  Difference in cerebral tissue oxygen saturation during sleep in patients with precapillary pulmonary hypertension at 2500m of high altitude with supplemental oxygen
Cerebral oxygen desaturation index without oxygen | 30 hours
  Difference in the cerebral oxygen desaturation index in patients with precapillary pulmonary hypertension at 2500m of high altitude without supplemental oxygen vs. low altitude
Cerebral oxygen desaturation index with oxygen | 30 hours
  Difference in the cerebral oxygen desaturation index in patients with precapillary pulmonary hypertension at 2500m of high altitude under supplemental oxygen.
Cerebral tissue oxygen saturation between different sleep stages | 30 hours
  Changes in the cerebral tissue oxygen saturation between different sleep stages at 2500 m compared to low altitude.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Lichtblau M, Schwarz EI, Ulrich T, Schneider SR, Bauer M, Furian M, Carta A, Forrer A, Saxer S, Muller J, Preiss H, Mayer L, Bloch KE, Ulrich S. Effect of an Overnight Stay at 2,500 Meters on Nocturnal Hypoxemia and Sleep-disordered Breathing in Patients with Pulmonary Vascular Disease: A Randomized Clinical Trial. Ann Am Thorac Soc. 2025 Jul;22(7):1053-1061. doi: 10.1513/AnnalsATS.202412-1279OC. PMID 40085143